CLINICAL TRIAL: NCT03194672
Title: Healthy Adolescent Transitions (HAT): A Comprehensive Approach to Targeting Adolescent Mothers
Brief Title: Healthy Adolescent Transitions (HAT)
Acronym: HAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jack Stevens (Other)
Collaborators: OhioHealth Research and Innovation Institute (Unknown)
Responsible Party: Sponsor-Investigator, Jack Stevens, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 90AP2678-01-00
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy Prevention; Life Skill Development

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Condition (Experimental): This experimental condition has three major components:
  1. Individual sessions: Roughly 12 90-minute sessions over 3 months Prenatal sessions covering contraceptive options, including long-acting reversible contraception. Prenatal and postnatal sessions will also cover (a) financial benefits of smoking cessation; (b)financial literacy/budgeting skills based upon selected components of the Money Matters curriculum; (c) establishing concrete steps to reach educational/career goals; (d) healthy eating habits; and (e) importance of HPV vaccinations and getting a medical home.
  2. Transportation assistance for medical home appointments.
  3. Electronic Prompts/Reminders to Encourage Completion of Goals.
  Interventions: Behavioral: Healthy Adolescent Transitions (HAT) program
- Treatment as Usual Control Condition (No Intervention): The comparison group will be a Usual Care control group. The control group will have access to standard medical and behavior health services as part of routine care. Prior to randomization, each enrolled participant will receive a listing of contact information for organizations offering this routine care.
  The only interaction the HAT providers will have with control group participants is to have periodic and brief phone conversations in which updated changes in contact information will be collected. The HAT providers will also obtain updated changes in contact information for HAT intervention group participants.

INTERVENTIONS:
Behavioral: Healthy Adolescent Transitions (HAT) program — The components of the intervention are described in the arm description.
  The intervention is based upon the theoretical framework of behavioral economics, which suggests that low intensity "nudges" can help recipients accomplish their own goals. All components of the intervention are voluntary; some participants may wish to discuss all components, while other participants may wish to discuss selected components consistent with their priorities.
  Arms: Intervention Condition

SUMMARY:
Randomized trial of a rapid repeat pregnancy prevention program for adolescent mothers.

Five hundred adolescent mothers from central Ohio will be enrolled--half will be assigned to an intervention that features nurses and social workers providing extra assistance during late pregnancy and the early postnatal period and half will be assigned to a standard of care intervention.

OhioHealth is the lead entity. Nationwide Children's Hospital serves as the local independent evaluator.

This federally funded contract is supported by the Family and Youth Services Bureau.

ELIGIBILITY:
Inclusion Criteria (at baseline)

1. Age 14-19 years
2. 24-35 weeks gestation
3. Medicaid insurance
4. Central Ohio resident
5. English speaking
6. Ability to provide informed consent (18-19 years of age) or minor assent and parental consent (<18 years of age)
7. Willingness to complete study-related surveys and coaching sessions
8. Patient must have her own smartphone, capable of running the study-related mobile application
9. Patient must have regular access to cellular or WiFi service

Exclusion Criteria

1. Patients < 13 years or >19 years
2. Non-English speaking
3. <24 or >35 weeks of gestation
4. Primary residence is located outside of central Ohio
5. Another adolescent from the household has already been enrolled in the program

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 331 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
Long acting reversible contraception | 12 months post enrollment
  Use of long acting reversible contraception
Repeat pregnancy | 21 months post enrollment
  Repeat pregnancy

SECONDARY OUTCOMES:
Nicotine use | 21 months post enrollment
  Use of cigarettes and vapor products
Financial literacy | 21 months post enrollment
  Understanding of financial terminology
School completion | 21 months post enrollment
  Highest grade completed
Medical home | 21 months post enrollment
  Use of primary care services
Healthy eating behaviors | 21 months post enrollment
  Eating nutritional food according to items from Youth Risk Behavior Survey
Employment | 21 months post enrollment
  Number of hours worked per week

CONTACTS AND LOCATIONS:
Overall Officials: Jack Stevens, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- OhioHealth Innovation Institute, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified data base will be available at conclusion of the study

REFERENCES:
- [Result] Stevens J, Rausch J, Osuagwu N, Lutz R. Efficacy of Behavioral Economic Nudges to Assist Teen Mothers: the Healthy Adolescent Transitions Randomized Controlled Trial. Prev Sci. 2024 Apr;25(3):509-520. doi: 10.1007/s11121-024-01660-3. Epub 2024 Mar 2. PMID 38429618